CLINICAL TRIAL: NCT04918160
Title: Evaluation of the Sanitary Safety of the French Intensive Care Society Annual Meeting Held From June 9th to June 11th 2021 at the Paris Congress Centre
Brief Title: Evaluation of the Sanitary Safety of a Healthcare Professional Conference Held 9-11 June 2021 in Paris
Acronym: COVID-FREE
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01185-36
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conference Attendees: Volunteering healthcare practitioners (medical doctor, nurse, nurse assistant, physiotherapist and psychotherapist) attending the FICS annual congress will be proposed to participate to the study.
  After giving their consent, participants will be asked to perform a COVID-19 antigenic screening self-test at day 7 (+/- 1) of the last day of the meeting (June 11th 2021) and to fill a questionnaire at day 21 of the last day of the meeting (June 11th 2021).
  Interventions: Other: Exposure to the FICS annual meeting (June 9-11 2021, Paris Congress Center)
- Controls: Volunteering healthcare practitioners (medical doctor, nurse, nurse assistant, physiotherapist and psychotherapist) not attending the FICS annual congress will be proposed to participate to the study. They will be recruited in the same medical departments as the Conference Attendees.
  After giving their consent, controls will be asked to perform a COVID-19 antigenic screening self-test at day 7 (+/- 1) of the last day of the meeting (June 11th 2021) and to fill a questionnaire at day 21 of the last day of the meeting (June 11th 2021).
  Interventions: Other: Exposure to the FICS annual meeting (June 9-11 2021, Paris Congress Center)

INTERVENTIONS:
Other: Exposure to the FICS annual meeting (June 9-11 2021, Paris Congress Center) — The study will compare COVID-19 screening nasal antigenic self-test (Boiron Auto Test Covid Nasal) positivity at D7 and COVID-19 symptoms in the 21 days between participants to the FICS annual meeting held in June 9-11 2021 in the Paris Congress Center (conference attendees / exposed) and healthcare professionals who did not attend the meeting (controls / not exposed).

SUMMARY:
The COVID-SRLF study will evaluate the sanitary safety of the French Intensive Care Society (FICS) annual meeting held in Paris Congress Center from June 9th to June 11th 2021 in the Coronavirus Disease 2019 (COVID-2019) pandemic situation. The primary objective is to determine the proportion of attendees with a positive antigenic COVID-19 screening test at day 7 (+/- 1) of their participation to the meeting. This rate will be compared to a cohort of health care professionals (medical doctors and paramedical professionals) from the same hospital ward as the attendees but who did not attend the meeting (stratified on centers, gender, age (< and >= 40 years, vaccination status (0, 1 or 2 doses) and socio-professional status (medical doctor, nurse, nurse assistant).

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professional healthy volunteer
* Absence of COVID-19 symptoms in the 2 weeks prior to inclusion
* Not being a COVID-19 contact case in the 2 weeks prior to inclusion
* Participation to at least one day of the FICS annual meeting (June 9-11 2021)

Exclusion Criteria:

* Non-healthcare professional (exhibitors, congress center employees)
* Refusal to participate to the study
* Person under legal protection
* Absence of social security affiliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two cohorts of healthy volunteers will be followed during 21 days after the French Intensive Care Society annual meeting. A first cohort, Conference Attendees cohort, constituted of volunteering healthcare practitioners (medical doctor, nurse, nurse assistant, physiotherapist and psychotherapist) attending the FICS annual congress. The second cohort, Control cohort, will gather volunteering healthcare practitioners (medical doctor, nurse, nurse assistant, physiotherapist and psychotherapist) who dit not attend the FICS annual congress, recruited in the same medical departments as the Conference Attendees participants.
Sampling Method: Non-Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Conference attendees COVID-19 prevalence at D7 | Day 7 of the last day of the meeting (June 18th, 2021)
  Proportion of conference attendees with a positive COVID-19 autotest at day 7 of the last day of the meeting (June 18th, 2021).

SECONDARY OUTCOMES:
Controls COVID-19 prevalence at D7 | Day 7 of the last day of the meeting (June 18th, 2021)
  Proportion of controls (healthcare professional not participating to the conference) with a positive COVID-19 autotest at day 7 of the last day of the meeting (June 18th, 2021).
Proportion of conference attendees with COVID-19 symptoms at D21 | Day 21 of the last day of the congress (July 2, 2021)
  Proportion of conference attendees reporting COVID-19 compatible symptoms until day 21 of the last day of the congress (July 2, 2021).
Proportion of conference attendees with COVID-19-related medical consultation at D21 | Day 21 of the last day of the congress (July 2, 2021)
  Proportion of conference attendees reporting COVID-19-related medical consultation until day 21 of the last day of the congress (July 2, 2021).
Proportion of conference attendees with COVID-19-related emergency department visit at D21 | Day 21 of the last day of the congress (July 2, 2021)
  Proportion of conference attendees reporting COVID-19-related emergency department visit until day 21 of the last day of the congress (July 2, 2021).
Proportion of conference attendees with COVID-19-related hospitalisation at D21 | Day 21 of the last day of the congress (July 2, 2021)
  Proportion of conference attendees reporting COVID-19-related hospitalisation until day 21 of the last day of the congress (July 2, 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Maury, MD, PhD, Principal Investigator — French Society for Intensive Care
Locations (1):
- Centre des Congres, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] SRLF Trial Group. Sanitary safety of the 2021 French Intensive Care Society medical conference: a case/control study. Ann Intensive Care. 2022 Feb 11;12(1):11. doi: 10.1186/s13613-022-00986-x. PMID 35147794